CLINICAL TRIAL: NCT01118013
Title: Reduced-Intensity Allogeneic Hematopoietic Cell Transplantation as Second Transplantation for Patients With Disease Relapse or Myelodysplasia After Prior Autologous Transplantation
Brief Title: Donor Stem Cell Transplant in Treating Patients With Relapsed Hematologic Malignancies or Secondary Myelodysplasia Previously Treated With High-Dose Chemotherapy and Autologous Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-100601; CALGB-100601; CDR0000667954 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); juvenile myelomonocytic leukemia; prolymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; recurrent adult Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; childhood diffuse large cell lymphoma; childhood grade III lymphomatoid granulomatosis; childhood immunoblastic large cell lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; post-transplant lymphoproliferative disorder; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes; recurrent childhood anaplastic large cell lymphoma; adult acute myelomonocytic leukemia (M4); childhood acute myelomonocytic leukemia (M4); adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); childhood acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); childhood acute promyelocytic leukemia (M3); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); childhood acute erythroleukemia (M6); adult acute megakaryoblastic leukemia (M7); childhood acute megakaryocytic leukemia (M7); childhood Burkitt lymphoma; atypical chronic myeloid leukemia, BCR-ABL1 negative; chronic myelomonocytic leukemia; cutaneous B-cell non-Hodgkin lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Leukemia, Myelomonocytic, Juvenile; Leukemia, Prolymphocytic; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Recurrence; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders | interventions — Antilymphocyte Serum; Filgrastim; Busulfan; fludarabine phosphate; Methotrexate; Mycophenolic Acid; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Matched-unrelated donor: Patients receive antithymocyte globulin, tacrolimus, and methotrexate as in HLA-identical donor regimen. Patients also receive oral mycophenolate mofetil twice daily on days 0 to 60.
  Allogeneic Stem Cell Transplantation: Patients undergo allogeneic peripheral blood stem cell transplantation on days 0 and 1. Patients then receive filgrastim subcutaneously daily beginning on day 7 and continuing until blood counts recover.
  Donor Lymphocyte Infusion (DLI): After day 180 (or day 210 for patients without an HLA-identical donor), patients with stable or progressive disease and no active GVHD may receive up to 3 DLIs every 8 weeks.
  Blood samples are collected at baseline and then periodically during study therapy for pharmacokinetic studies.
  After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for up to 5½ years.
  Interventions: Biological: anti-thymocyte globulin; Biological: donor lymphocytes; Biological: filgrastim; Biological: therapeutic allogeneic lymphocytes; Drug: busulfan; Drug: fludarabine phosphate; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: tacrolimus; Other: reduced-intensity transplant conditioning procedure; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: donor lymphocytes
Biological: filgrastim
Biological: therapeutic allogeneic lymphocytes
Drug: busulfan
Drug: fludarabine phosphate
Drug: methotrexate
Drug: mycophenolate mofetil
Drug: tacrolimus
Other: reduced-intensity transplant conditioning procedure
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy, such as busulfan and fludarabine phosphate, before a peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving methotrexate, tacrolimus, and antithymocyte globulin before and after the transplant may stop this from happening. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer cells as not belonging in the patient's body and destroy them (called graft-versus-tumor effect). Giving an infusion of the donor's white blood cells (donor lymphocyte infusion) may boost this effect.

PURPOSE: This phase II trial is studying how well donor stem cell transplant works in treating patients with relapsed hematologic malignancies or secondary myelodysplasia previously treated with high-dose chemotherapy and autologous stem cell transplant .

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To demonstrate the efficacy of performing reduced-intensity conditioning allogeneic hematopoietic cell transplantation in patients with relapsed hematologic malignancies or secondary myelodysplasia after completion of prior high-dose chemotherapy and autologous hematopoietic stem cell transplantation.
* To compare the strategy of this regimen with the strategy used in CALGB-100002.

Secondary

* To describe the response rate at 6 and 12 months in patients treated with this regimen.
* To describe the time-to-progression in patients treated with this regimen.
* To determine the ability to use pharmacokinetic-directed busulfan to achieve AUC within 20% of target AUC in > 80% of patients.
* To determine percent of donor chimerism in T-cell, myeloid and B-cell populations achieved with this regimen compared with CALGB-100002.
* To determine the risk of acute and chronic graft-versus-host disease and other toxicities of this regimen in these patients.
* To describe the overall survival and disease-free survival of patients treated on this regimen.
* To determine the rate of viral, bacterial, and fungal opportunistic infections occurring in the first year after transplantation compared with CALGB-100002.

OUTLINE: This is a multicenter study.

* Preparative Regimen:

  * Busulfan test dose: Patients receive busulfan IV over 45 minutes once during days -14 and -9.
  * Busulfan treatment dose: Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -3 and busulfan IV over 3 hours on days -6 to -3.
* Graft-vs-Host Disease (GVHD) Prophylaxis:

  * HLA-identical donor: Patients receive antithymocyte globulin IV over 6-10 hours on days -6 to -5; oral tacrolimus twice daily on days -2 to 90 followed by a taper* as tolerated until day 150 or 180; and methotrexate IV on days 1, 3, and 6.

NOTE: * Tacrolimus may be tapered on days 60-90 if donor chimerism of CD3+ cells is < 50% at day 60 or patient has progressive disease.

* Matched-unrelated donor: Patients receive antithymocyte globulin, tacrolimus, and methotrexate as in HLA-identical donor regimen. Patients also receive oral mycophenolate mofetil twice daily on days 0 to 60.

  * Allogeneic Stem Cell Transplantation: Patients undergo allogeneic peripheral blood stem cell transplantation on days 0 and 1. Patients then receive filgrastim subcutaneously daily beginning on day 7 and continuing until blood counts recover.
  * Donor Lymphocyte Infusion (DLI): After day 180 (or day 210 for patients without an HLA-identical donor), patients with stable or progressive disease and no active GVHD may receive up to 3 DLIs every 8 weeks.

Blood samples are collected at baseline and then periodically during study therapy for pharmacokinetic studies.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for up to 5½ years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hematologic malignancies:

  * Chronic lymphocytic leukemia (CLL) or prolymphocytic leukemia (PLL)

    * Absolute lymphocytosis of > 5,000/μL
    * Lymphocytes must appear morphologically mature with < 55% prolymphocytes (CLL)

      * Patients with > 55% prolymphocytes are considered as having PLL
    * Lymphocyte phenotype with expression of CD20, CD19, and CD5 (CLL)
  * Non-Hodgkin lymphoma

    * Any WHO classification of histologic subtype
    * Core biopsies acceptable for primary diagnosis and immunophenotyping
    * Bone marrow biopsies as sole means of diagnosis not allowed for follicular lymphoma
  * Hodgkin lymphoma

    * Any WHO classification of histologic subtype
    * Core biopsies acceptable for primary diagnosis and immunophenotyping
    * Bone marrow biopsy is required
  * Multiple myeloma

    * Patients must have active disease requiring treatment (Durie-Salmon stage I-III)
  * Acute myeloid leukemia

    * Must have < 10% bone marrow blasts and no circulating blasts
  * Myelodysplastic syndrome (MDS)

    * MDS as define by WHO criteria
    * Must have < 10% marrow blasts
* Relapsed or progressive disease or myelodysplasia ≥ 6 months after prior high-dose chemotherapy with autologous hematopoietic cell support

  * Prior syngeneic transplantation allowed
* Healthy donor meeting one of the following criteria:

  * HLA-identical sibling (6/6)

    * Serologic typing for class I (A, B) and molecular typing for class II (DRB1) required
  * 8/8 matched-unrelated donor

    * Molecular identity at HLA A, B, C, and DRB1 by high-resolution typing required
  * No syngeneic donors

PATIENT CHARACTERISTICS:

* Creatinine clearance ≥ 40 mL/min
* Total bilirubin ≤ 2 mg/dL
* AST ≤ 3 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* DLCO ≥ 40% with no symptomatic pulmonary disease
* LVEF ≥ 30% by MUGA or ECHO
* No uncontrolled diabetes mellitus or active serious infection
* No known hypersensitivity to E.coli-derived products
* No HIV infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks should elapse between prior standard cytotoxic chemotherapy, radiation therapy, or surgery and the planned start of the preparative regimen on day -7

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asad Bashey, MD, PhD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (10):
- United States (10):
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton MD, Maryland
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2010 and March 2012, 6 participants were recruited.
Groups:
- Treatment: Participants will receive:
  Busulfan test dose of 25 mg/m^2 IV over 45 minutes between days -14 and -9; Fludarabine 30 mg/m^2/day IV over 30 minutes on days -7 to -3; Busulfan IV x 4 days on days -6 through -3 (dosage based on AUC of 4000 mmol/min based on pharmacokinetics determined from test dose); Allopurinol was given at discretion of treating physician; Rabbit antithymocyte globulin 1.5 mg/kg/day IV on days -6 and -5; Peripheral Blood Stem Cell Transplant (PBST) on Day 0 and +1; and methotrexate 5 mg/m^2/day IV on days +1, +3 and +6. G-CSF of 5mcg/kg/day SQ began daily on day +7 continuing until ANC > 1000/mL for 3 consecutive days.
Period: Overall Study
Arm/Group | Treatment
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 67 [58 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: EFS was defined as the date of transplant to date of progression or develop myelodysplasia after autologous transplant. EFS was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 5.5 years)
Population: Due to study termination, data were not collected and the outcome measure was not analyzed.
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Primary Outcome: Comparison of EFS Distribution to That of CALGB-100002
Description: EFS distributions between CALGB-100002 and this study will be compared using the two-sample log-rank test.
Time Frame: 2 years
Population: Due to study termination, data were not collected and the outcome measure was not analyzed.
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Complete Response Rate
Description: Complete response (CR) rate is reported as the percentage of participants who achieved a CR.
Time Frame: Up to 5.5 years
Population: Due to study termination, data were not collected and the outcome measure was not analyzed.
Arm/Group | Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the transplant from registration to death of any cause. Surviving patients were censored at the date of last follow-up. The median OS with 95% confidence interval (CI) was estimated using the Kaplan Meier method.
Time Frame: Up to 5.5 years
Population: Due to study termination, data were not collected and the outcome measure was not analyzed.
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Rate of Opportunistic Infections
Description: Percent of participants who have an opportunistic (viral, bacterial and fungal) infection in the first year following transplant.
Time Frame: 1 year post transplant
Population: Due to study termination, data were not collected and the outcome measure was not analyzed.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Flashing lights (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=6)
Anemia (Blood and lymphatic system disorders) | 6 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (3)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (2)
Watering eyes (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 4 (7)
Dry mouth (Gastrointestinal disorders) | 3 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 3 (6)
Oral pain (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (5)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 3 (4)
Fatigue (General disorders) | 4 (12)
Fever (General disorders) | 3 (8)
Pain (General disorders) | 2 (3)
Catheter related infection (Infections and infestations) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 3 (7)
Lung infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (13)
Alkaline phosphatase increased (Investigations) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 5 (13)
Blood bilirubin increased (Investigations) | 2 (2)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 6 (16)
GGT increased (Investigations) | 1 (1)
INR increased (Investigations) | 2 (2)
Investigations - Other, specify (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (13)
Platelet count decreased (Investigations) | 6 (18)
Weight loss (Investigations) | 4 (5)
White blood cell decreased (Investigations) | 2 (8)
Anorexia (Metabolism and nutrition disorders) | 4 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (7)
Hypokalemia (Metabolism and nutrition disorders) | 2 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (6)
Hyponatremia (Metabolism and nutrition disorders) | 4 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (3)
Dysgeusia (Nervous system disorders) | 2 (4)
Headache (Nervous system disorders) | 1 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (4)
Insomnia (Psychiatric disorders) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (9)
Hypotension (Vascular disorders) | 4 (6)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less